CLINICAL TRIAL: NCT03033004
Title: Cryolipolisis for Subcutaneous Abodomen and Flank Fat Reduction
Brief Title: Cryolipolisis for Abdomen and Flank Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Richard Eloin Liebano, PT, PhD, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 61499416.5.0000.5490
Record Dates: First submitted 2017-01-10; First posted 2017-01-26 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Subcutaneous Fat Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional Cryolipolysis (Active Comparator): Subjects will receive one treatment session of conventional cryolipolisys. Subcutaneous fat tissue will be cooled with the cryolipolitic device for 60 minutes. The treatmente area will be the abdomen and/or flanks according to each patient's needs (pragmatic treatment).
  Interventions: Device: Conventional Cryolipolysis
- Contrast Cryolipolysis (Active Comparator): Subjects will receive one treatment session of contrast cryolipolisys. Subcutaneous fat tissue will be heated for 10 minutes, cooled for 60 minutes, and heated again for 10 minutes with the cryolipolitic device. The treatmente area will be the abdomen and/or flanks according to each patient's needs (pragmatic treatment).
  Interventions: Device: Contrast Cryolipolysis
- Reperfusion Cryolipolysis (Active Comparator): Subjects will receive one treatment session of Reperfusion Cryolipolysis. Subcutaneous fat tissue will be cooled with the cryolipolitic device for 60 minutes and heated for 10 minutes. The treatmente area will be the abdomen and/or flanks according to each patient's needs (pragmatic treatment).
  Interventions: Device: Reperfusion Cryolipolysis

INTERVENTIONS:
Device: Conventional Cryolipolysis — Treatment will be a cold exposure of the subcutaneous fat for 60 minutes using the Polarys device. Polarys is a commercially available cryolipolitic device.
  Arms: Conventional Cryolipolysis
Device: Contrast Cryolipolysis — Treatment will consist of a heat exposure of the subcutaneous fat for 10 minutes followed by 60 minutes of cold exposure and 10 minutes of heat exposure again. Cold and heat will be provided by the Polarys device. Polarys is a commercially available cryolipolitic device.
  Arms: Contrast Cryolipolysis
Device: Reperfusion Cryolipolysis — Treatment will be a cold exposure of the subcutaneous fat for 60 minutes followed by 10 minutes of heat exposure using the Polarys device. Polarys is a commercially available cryolipolitic device.
  Arms: Reperfusion Cryolipolysis

SUMMARY:
Sixty healthy subjects aged between 18 and 50 will be randomly allocated into three treatment groups: Conventional Cryolipolysis, Contrast Cryolipolysis or Recovery Reperfusion Cryolipolysis. The region will be treated according to the individual need, in the region of abdomen and flanks. Assessments of body composition will be performed at baseline and 30, 60 and 90 days after randomization. Blood collections will also be performed at baseline and between 14 and 21 days after randomization for evaluation of lipid profile and liver function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body mass index > 29.9 Kg/m2

Exclusion Criteria:

* Pregnancy
* Diabetes
* Cancer
* Vascular diseases
* Heart diseases
* Liposuction or other surgical procedures for body contouring
* Active infection
* Wounds
* Paroxysmal cold hemoglobinuria
* Cold urticaria
* Significant weight changes in the past 3 months or during treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Fat layer thickness changes measured by ultrasound | 90 days after randomization

SECONDARY OUTCOMES:
Fat layer thickness changes measured by ultrasound | 30 days after randomization
Fat layer thickness changes measured by ultrasound | 60 days after randomization
Changes in skin viscoelasticity measured by a cutometer | 30 days after randomization
Changes in skin viscoelasticity measured by a cutometer | 60 days after randomization
Changes in skin viscoelasticity measured by a cutometer | 90 days after randomization
Changes in cholesterol levels | 21 days after randomization
  Cholesterol levels will be measured in mg/dL
Changes in triglyceride levels | 21 days after randomization
  Triglyceride levels will be measured in mg/dL
Changes in blood levels of alanine aminotransferase (ALT) | 21 days after randomization
Changes in blood levels of aspartate transaminase (AST) | 21 days after randomization
Changes in fasting blood glucose | 21 days after randomization
Changes in circumference measurements | 30 days after randomization
Changes in circumference measurements | 60 days after randomization
Changes in circumference measurements | 90 days after randomization
Changes in body weight | 30 days after randomization
Changes in body weight | 60 days after randomization
Changes in body weight | 90 days after randomization
Subject's satisfaction with regard to treatment measued by a numeric scale ranging from 1 to 3. | 90 days after randomization
  1= unsatisfied; 2= indifferent; 3= satisfied
Subject's tolerance with regard to treatment measued by a numeric scale ranging from 1 to 3. | 90 days after randomization
  1 = intolerable; 2= tolerable; 3= comfortable

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Estudos e Formação Avançada Ibramed., Amparo, São Paulo, Brazil